CLINICAL TRIAL: NCT01453400
Title: Onset of Action of a Fast Release Aspirin Tablet and Acetaminophen Caplet in Sore Throat Pain
Brief Title: Evaluate the Time of Pain Relief of Fast Acting Aspirin Versus Acetaminophen in Subjects Diagnosed With Sore Throat Pain
Acronym: Tarot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15772
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Pharyngitis
Keywords: aspirin; acetylsalicylic acid; pharyngitis; sore throat
MeSH Terms: conditions — Pharyngitis | interventions — Aspirin; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAY1019036) + placebo
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetaminophen + placebo
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin, BAY1019036) + placebo — Single dose, 2 x 500 mg fast release aspirin tablets (1000 mg) + 2 x placebo acetaminophen caplets
  Arms: Arm 1
Drug: Acetaminophen + placebo — Single dose, 2 x 500 mg Acetaminophen caplets (1000 mg) + 2 x placebo fast release Aspirin tablets
  Arms: Arm 2
Drug: Placebo — Single dose, 2 x placebo Acetaminophen caplets + 2 x placebo fast release Aspirin tablets
  Arms: Arm 3

SUMMARY:
This study is to evaluate the onset of relief provided by a single, oral dose of fast release aspirin 1000 mg compared to acetaminophen 1000 mg and placebo in subjects with sore throat pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female subjects ≥ 18 years of age
* Presence of sore throat due to upper respiratory tract infection (URTI)
* Onset of sore throat pain within six days of the screening period
* Baseline sore throat pain intensity score ≥ 60 mm on the Sore Throat Pain Intensity Scale
* Have a score ≥ 5 on the Tonsillopharyngitis Assessment
* Female subjects of childbearing potential who are currently sexually active must be using a medically acceptable form of birth control for at least one month prior to screening (three months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, Nuvaring, Depo-Provera, or double-barrier and have a negative pregnancy test at screening/treatment period. Female subjects of non-childbearing potential must be amenorrheic for at least two years or had a hysterectomy and/or bilateral oophorectomy.
* Understand the pain rating assessments

Exclusion Criteria:

* History of hypersensitivity to aspirin, salicylates, other nonsteroidal anti-inflammatory drugs, acetaminophen, opioid analgesics, and similar drugs
* Use of any "cold medication" (i.e. decongestants, antihistamines, expectorants, antitussives) within four hours preceding administration of the investigational product
* Use of any immediate release analgesic/antipyretic within four hours or use of any sustained release or long-acting analgesic/antipyretic within twelve hours preceding administration of the investigational product
* Consumption of alcoholic beverages, or foods and beverages containing xanthines within two hours prior to administration of the investigational product
* Use of any sore throat lozenges, sprays, cough drops, menthol-containing products within one hour preceding administration of the investigational product
* Presence of cough that causes throat discomfort
* Presence of mouth-breathing or any respiratory condition that, in the Investigator's judgment, could compromise breathing
* Evidence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies for which aspirin or acetaminophen is contraindicated
* Relevant concomitant disease such as medically uncontrolled asthma (exercise induced asthma is permitted), chronic sinusitis or nasal structural abnormalities causing greater than fifty percent obstruction
* History of gastrointestinal bleeding or perforation related to previous non-steroidal anti-inflammatory therapy.
* Current or past history of a bleeding disorder
* Self reported alcoholism or drug abuse within two years prior to screening or routine consumption of three or more alcohol containing beverages per day
* Habituation to analgesic drugs or tranquilizers (i.e., routine use of five or more times per week for greater than three weeks)
* Acute illness, local infection, or disease (other than URTI with pharyngeal infection) that can interfere with the conduct of the study
* Current use of blood thinning (anticoagulant), low dose aspirin, or steroid drug
* Has initiated treatment for depression within the past thirty days
* Females who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2011-09-27 (Actual); Primary Completion 2012-04-05 (Actual); Study Completion 2012-04-06 (Actual)

PRIMARY OUTCOMES:
Time to meaningful pain relief from the Sore Throat Pain Intensity Scale (STPIS) 100 mm visual analog scale | Up to two hours

SECONDARY OUTCOMES:
Global assessment of the investigational product as a pain reliever by grading from 0 to 4 (from poor to excellent) | Two hours postdose or immediately before the intake of rescue medication
Time to first perceptible relief (defined as the time when the subject presses the first stopwatch) | Up to two hours
Time weighted sum of pain intensity differences (PID) scores over first hour | Up to one hour
Time weighted sum of pain intensity differences (PID) scores over 2 hours | Up to two hours
Percentage difference from baseline Sore Throat Pain Intensity Scale (STPIS) to STPIS at time of meaningful relief | Up to two hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Storrs, Connecticut, United States

REFERENCES:
- [Derived] Voelker M, Schachtel BP, Cooper SA, Gatoulis SC. Efficacy of disintegrating aspirin in two different models for acute mild-to-moderate pain: sore throat pain and dental pain. Inflammopharmacology. 2016 Feb;24(1):43-51. doi: 10.1007/s10787-015-0253-0. Epub 2015 Nov 24. PMID 26603742